CLINICAL TRIAL: NCT07325396
Title: Effectiveness of Neuromuscular Training Added to Routine Practice on Fatigue and Stress Biomarkers in Professional Esports Players: A Randomized Controlled Trial
Brief Title: Neuromuscular Training in Professional Esports Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Doğukan Tongar, Teaching Assistant, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-SPORT-NME-2025-01
Record Dates: First submitted 2025-11-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Esports; Esports Players
Keywords: esports; professional gamers; neuromuscular training; fatigue; stress; biomarkers
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training (Experimental): Professional esports players will perform a structured neuromuscular training program added to their routine esports practice, 3 sessions per week for 8 weeks. The program includes warm-up, aerobic, strengthening, core stabilization, functional and reaction drills with progressive weekly increases in duration or repetitions.
  Interventions: Behavioral: Neuromuscular Training
- Physical Activity Counseling (Active Comparator): Professional esports players will receive structured physical activity counseling in addition to their routine esports practice. The counseling will follow ACSM 5A principles (Assess, Advise, Agree, Assist, Arrange) to support behavior change and increase physical activity participation weekly for 8 weeks.
  Interventions: Behavioral: Physical Activity Counseling

INTERVENTIONS:
Behavioral: Neuromuscular Training — A progressive neuromuscular exercise program including dynamic warm-up, aerobic exercises, functional strengthening of lower and upper extremity muscles, core stabilization training, and reaction drills performed 3 times per week for 8 weeks. Duration and repetitions increase biweekly according to a structured progression protocol.
  Arms: Neuromuscular Training
Behavioral: Physical Activity Counseling — Structured physical activity counseling based on ACSM 5A principles (Assess, Advise, Agree, Assist, Arrange) delivered weekly for 8 weeks to promote sustainable physical activity behaviors and reduce sedentary time during esports training routines.
  Arms: Physical Activity Counseling

SUMMARY:
Professional esports players engage in prolonged training sessions and experience high physical and mental stress due to intensive competition schedules. These demands can lead to increased fatigue, decreased performance, and health problems. This randomized controlled trial aims to investigate whether adding a structured neuromuscular exercise program to routine esports training reduces fatigue and stress biomarkers and improves performance-related outcomes in professional esports players.

DETAILED DESCRIPTION:
Esports players often perform long hours of training that require sustained physical and cognitive effort, which may result in musculoskeletal problems, mental fatigue, and elevated stress levels. Most studies in the esports field rely on subjective evaluations and include non-professional populations. Objective assessment of fatigue and stress biomarkers in professional esports athletes is still lacking.

This prospective randomized controlled trial will include 24 professional esports players aged 18-35 who train at least 35 hours per week with their teams. Participants will be randomly assigned to either a neuromuscular training group or a control group. The intervention group will complete an 8-week neuromuscular exercise program three times per week in addition to their regular esports training routine. The control group will receive structured physical activity counseling based on ACSM 5A principles.

Primary outcomes include serum levels of cortisol, testosterone, testosterone/cortisol ratio, C-reactive protein (CRP), creatine kinase (CK), vitamin B12, and iron measured under standardized fasting conditions. Secondary outcomes include muscle strength (myometry), sleep quality (Pittsburgh Sleep Quality Index), physical activity level (IPAQ-SF), quality of life (SF-12), visual and auditory reaction time tests, lactate measures (Lactate Scout), and mood states (POMS). Outcomes will be assessed at baseline and after the 8-week intervention period.

The findings of this study are expected to provide evidence-based recommendations for integrating neuromuscular conditioning into professional esports training to enhance physical health, reduce fatigue and stress, and improve overall performance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 years
* Currently competing as a contracted professional esports player
* Playing one of the following games at a professional level:

League of Legends, Counter Strike 2, Overwatch, Valorant, Apex Legends, DOTA2, Rocket League, PUBG

* Participating in ≥35 hours/week of training with their team
* Voluntary agreement to participate and sign informed consent

Exclusion Criteria:

* History or presence of medical conditions affecting safety or performance: metabolic, cardiovascular, renal, neurological, or respiratory disorders

  * Playing esports only at amateur or beginner level
  * Answering "Yes" to any item in the Physical Activity Readiness Questionnaire (PAR-Q)

Removal Criteria:

* Participating in <35 hours/week esports training during the study
* Missing ≥2 neuromuscular training sessions (intervention group)
* Leaving their professional esports organization (roster removal, retirement, etc.)
* Any illness or injury preventing continuation of esports participation

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum cortisol level - Stress Biomarkers | Baseline and 8 weeks
  Serum cortisol level will be analyzed under fasting conditions using standardized laboratory protocols.
Testosterone level - Stress Biomarkers | Baseline and 8 weeks
  Testosterone level will be analyzed under fasting conditions using standardized laboratory protocols.
C-Reactive Protein Level (CRP) - Fatigue Biomarkers | Baseline and 8 weeks
  Serum CRP levels will be analyzed under fasting conditions using standardized laboratory protocols.
Creatine Kinase (CK) Level - Fatigue Biomarkers | Baseline and 8 weeks.
  Creatine kinase levels will be analyzed under fasting conditions using standardized laboratory protocols.
Vitamin B12 Level - Fatigue Biomarkers | Baseline and 8 weeks.
  Serum vitamin B12 levels will be analyzed under fasting conditions using standardized laboratory protocols.
Iron Level - Fatigue Biomarkers | Baseline and 8 weeks.
  Serum iron levels will be analyzed under fasting conditions using standardized laboratory protocols.

SECONDARY OUTCOMES:
Muscle Strength | Baseline and 8 weeks
  Hand, forearm, shoulder, and back muscle strength will be assessed using a handheld myometer; mean of three trials recorded in kilograms.
Sleep Quality | Baseline and 8 weeks
  Assessment of subjective sleep quality, sleep duration, sleep disturbances, and overall sleep efficiency with Pittsburgh Sleep Quality Index.
  The Pittsburgh Sleep Quality Index (PSQI) consists of 19 items that generate seven component scores, each ranging from 0 to 3, yielding a global score between 0 and 21, with higher scores indicating poorer sleep quality; a total score greater than 5 reflects clinically significant sleep disturbance.
Physical Activity Level | Baseline and 8 weeks
  Self-reported physical activity levels converted to MET-minutes per week. (IPAQ-Short Form). The International Physical Activity Questionnaire-Short Form (IPAQ-SF) provides total physical activity expressed in Metabolic Equivalent of Task (MET)-minutes/week, and scores are categorized as follows: <600 MET-minutes/week indicates low activity, 600-3000 MET-minutes/week indicates moderate activity, and >3000 MET-minutes/week indicates high physical activity level.
Reaction Time | Baseline and 8 weeks
  Average visual reaction time over 5 trials recorded in milliseconds. Average response latency to an auditory stimulus over 5 trials.
Blood Lactate Concentration | Baseline and 8 weeks
  Capillary blood lactate measured to assess metabolic response to neuromuscular training.
Mood State | Baseline and 8 weeks
  Assessment of tension, depression, anger, fatigue, and vigor subscales with Profile of Mood States (POMS). The Profile of Mood States (POMS) assesses mood across multiple dimensions and yields a Total Mood Disturbance (TMD) score by summing negative mood subscales and subtracting the vigor score; higher TMD scores indicate greater mood disturbance, whereas lower scores reflect better overall mood.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy protection and confidentiality regulations for professional esports players.

REFERENCES:
- [Background] Ambrozy T, Rydzik L, Obminski Z, Blach W, Serafin N, Blach B, Jaszczur-Nowicki J, Ozimek M. The Effect of High-Intensity Interval Training Periods on Morning Serum Testosterone and Cortisol Levels and Physical Fitness in Men Aged 35-40 Years. J Clin Med. 2021 May 15;10(10):2143. doi: 10.3390/jcm10102143. PMID 34063524
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Andre TL, Walsh SM, ValladAo S, Cox D. Physiological and Perceptual Response to a Live Collegiate Esports Tournament. Int J Exerc Sci. 2020 Sep 1;13(6):1418-1429. doi: 10.70252/KNEB6696. eCollection 2020. PMID 33042382
- [Background] Nagorsky E, Wiemeyer J. The structure of performance and training in esports. PLoS One. 2020 Aug 25;15(8):e0237584. doi: 10.1371/journal.pone.0237584. eCollection 2020. PMID 32841263
- [Background] Bonnar D, Castine B, Kakoschke N, Sharp G. Sleep and performance in Eathletes: for the win! Sleep Health. 2019 Dec;5(6):647-650. doi: 10.1016/j.sleh.2019.06.007. Epub 2019 Jul 15. PMID 31320292
- [Background] Emara AK, Ng MK, Cruickshank JA, Kampert MW, Piuzzi NS, Schaffer JL, King D. Gamer's Health Guide: Optimizing Performance, Recognizing Hazards, and Promoting Wellness in Esports. Curr Sports Med Rep. 2020 Dec;19(12):537-545. doi: 10.1249/JSR.0000000000000787. PMID 33306517
- [Background] DiFrancisco-Donoghue J, Balentine J, Schmidt G, Zwibel H. Managing the health of the eSport athlete: an integrated health management model. BMJ Open Sport Exerc Med. 2019 Jan 10;5(1):e000467. doi: 10.1136/bmjsem-2018-000467. eCollection 2019. PMID 30792883
- [Background] Jenny, S. E., Manning, R. D., Keiper, M. C., & Olrich, T. W. (2017). Virtual (ly) athletes: where eSports fit within the definition of "Sport". Quest, 69(1), 1-18.